CLINICAL TRIAL: NCT02948491
Title: Effectiveness of Music Therapy on the Intra-hospital Evolution and Neurodevelopment of Preterm Neonates Treated in Neonatal Intensive Care Units in the Bucaramanga Metropolitan Area
Brief Title: Effectiveness of Music Therapy on the Development of Preterm Neonates
Acronym: EMT-DRNP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Manuela Beltrán (Other)
Collaborators: Fundación Cardiovascular de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2016-10-18; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Premature Birth
Keywords: Complementary Therapies; Neonate Intensive Care Units (NICU); Child Development; Infants Premature
MeSH Terms: conditions — Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music therapy (Experimental): First. Recording of the voice of the mother singing the song to the child. (To choose this option, the song must be sung to the child during pregnancy at least 2 to 3 times per week. Second. The mother's favorite song, obtained externally. (To choose this option, the mother must bring the song that she that she listened to frequently, at least 5 times per week). Third. Pre-determined lullaby. (This option refers only to the lullaby melody or Brahms lullaby, edited to obtain stable volumes and normalization of the audio, with the effect of progressively appearing and fading for the first and last 10 seconds of the intervention with music therapy, so there are no drastic acoustic changes in the intervention. Audacity editing software will be used.)
  Interventions: Other: Music therapy
- Without sound emission (No Intervention): The infant does not receive any sound emission because the baffle will be turned off.
  One of the three "intervention" options are chosen. The parents are told that their child may be randomly assigned to either the therapeutic or control group.

INTERVENTIONS:
Other: Music therapy — Song that the mother sings to the child before birth, recording of the mother's voice.
  Arms: Music therapy

SUMMARY:
Pragmatic, randomized controlled clinical trial with blinding of the evaluator, performed in order to estimate the effectiveness, six (6) months after hospital discharge, of music therapy on the intra-hospital evolution and neurodevelopment of preterm neonates (gestational ages 28 to 37weeks) who are treated in Neonatal Intensive Care Units (NICU) in the Bucaramanga Metropolitan Area.

DETAILED DESCRIPTION:
This is a pragmatic, randomized controlled clinical trial with blinding of the evaluator, performed in order to estimate the effectiveness, six (6) months after hospital discharge, of music therapy on the intra-hospital evolution and neurodevelopment of preterm neonates (gestational ages 28 to 37weeks) who are treated in Neonatal Intensive Care Units (NICU) in the Bucaramanga Metropolitan Area.

The study population is premature neonates at gestational ages 28 to 37 weeks who are treated in Neonatal Intensive Care Units (NICU). They will receive an intra-hospital music therapy intervention and will be compared to premature neonates in the same unit who will receive an intervention without sound emissions. The purpose is to identify differences in the behavior of clinical parameters at the intra-hospital level as well as in neurodevelopment six (6) months after hospitalization.

To begin recruitment for the study, a neonatologist will contact the father/mother or legal representative and will briefly explain the purpose of the study and its procedures. After this, if the father/mother or legal representative is interested in allowing the neonate to participate, they will be put in contact with the physiotherapist coordinating the study who will fully explain the research. The neonate's participation in the study will be confirmed by an informed consent form signed by the parents. Each subject will be randomly assigned to an intervention group (music therapy or no sound emissions) based on a previously generated random numbers table. The person who possesses this table will indicate to the project coordinator via telephone the group to which each neonate is assigned, which will be stratified according to the healthcare clinic.

Since this is a pragmatic trial, given the nature of the intervention, before the trial the mother will need to decide which of three music therapy options she would like her child to receive: her favorite song which she will sing, her favorite song which is obtained externally or a lullaby. This process of choosing the song is done only when assigned to the music therapy group, but the parents or legal representative will be told that their child could be assigned to either of the two groups, with music therapy or without sound emissions. At no time during the interventions will the parents, representative or the health professionals know the group to which the preterm neonate is assigned.

The intervention will begin 24 hours after birth or when admitted to the clinic and will start by collecting the data requested on the admissions form. The sample will be composed of 90 neonates, 45 of which will receive music therapy and 45 will receive intervention without sound emissions. This sample was estimated based on an alpha of 0.05 and a power of 0.9.

The intervention parameters for volume intensity will be 55-65 decibels (db). The intervention will be performed by two physiotherapists who will alternate shifts to cover all the intervention days, since these two people will carry out the intervention on all of the days during which the infants will remain hospitalized. The exposure time will be 15 minutes per day. A mini baffle (JBL Bluetooth Go Brand) will be individually placed in a sealed sterile sleeve and put inside the incubator or on the top-center part of the crib aligned with the head of the neonate. The decibels will be measured with a Sonometer, which will be placed on the edge of the top access window on the right side of the incubator, facing in the direction of the neonate's ear.

The variables to be registered for each intervention are: heart rate, respiratory rate, oxygen saturation and blood pressure. Each variable will be measured before the intervention, at 5, 10 and 15 minutes into the intervention, and 5 minutes after the intervention. During this time, the infant will be observed and any physical changes will be registered, including movement, crying, calming or anything that is different from the ordinary daily development of the neonate. When the infant is discharged (either to the pediatric intensive/intermediate care unit or home), a discharge report will be completed which will describe the clinical conditions under which the infant is leaving the unit. If the infant continues to be hospitalized in another unit, such as the pediatric/intermediate unit, he or she will receive the intervention until leaving the clinic, with the same parameters mentioned previously.

In addition, a nurse in each unit (neonatal or pediatric) will register the changes from the previous day using a clinical monitoring data collection form, which includes the variables: relevant changes in vital signs, diagnoses, treatments, etc. (information obtained from the clinical chart or from the printed nursing report).

All the measurement procedures will be standardized prior to application. The evaluators will be trained in the field using a pilot test, based on which the needed corrections will be applied. In addition, 10% of the measurements will be repeated or verified by the field coordinator. All the evaluators will be blinded to the intervention assignments and to the clinical status of the patients in order to prevent differential information bias.

The father/mother, legal representative or medical team can decide to withdraw the infant from the study at any time and for any reasons they consider valid. The reason for withdrawal will be recorded on the last monitoring form that is completed.

If the infant is discharged and on the next day is again hospitalized, and the Bayley III evaluation of the development of the infant has not yet been obtained, he or she will continue to receive the intervention in the hospital according to the protocol described by this study. If the Bayley III evaluation has been obtained and the infant returns to the clinic, the infant will not be treated because he or she would already be part of the next phase of the study, which involves the neurodevelopment of the infant.

When the infant meets the criteria (corrected developmental age and is not hospitalized), the researcher shall immediately contact the father/mother or legal representative to perform a Bayley III evaluation of the development of the infant, which must be performed no later than six (6) days post-hospitalization. This evaluation will be conducted in the laboratories of the Manuela Beltran University (Gesell campus) under the following parameters: the evaluators (psychologist and physiotherapist) shall have at least 6 months of prior experience working with infants and will be trained in the use of this development scale prior to its application; the evaluators will be blinded to the type of intervention the infant is receiving; the evaluations (psychological and physiotherapeutic) will be performed simultaneously and the professionals will not be able to communicate among themselves during the intervention, and they will be recorded and monitored in order to ensure this condition is met; in addition, with no prior warning, the project coordinator will periodically monitor the evaluators through a one-way mirror located in the laboratory. The evaluators will electronically record the data on two laptop computers (using Bayley III software) located far away from each other in the laboratory, and will give an electronic and printed copy of the Bayley III evaluation form to the coordinator before leaving the laboratory. The two types of registries must agree, which will serve as a strategy to control the quality of the data. This evaluation will be repeated six months after hospitalization under the same conditions and by the same evaluators.

During the first six months after hospitalization, the coordinator will call the parents or legal representative every 15 days, with four objectives: achieve adherence to the project, update contact data, identify the health conditions of the infant; and remind the parents or legal representative of the different check-ups that the child should receive during those six months.

To this end, a general follow-up form will exist, which will contain the personal data of the infant and the father/mother or legal representative, the intensive care unit where he or she is treated, situations pertinent to the infant's condition, review of the dates of the post-hospitalization follow-up calls; review of completion of daily nursing forms, interventions, the 2 Bayley III evaluations, among others, in order to generate a database and to collect the data at the times established.

To handle missing data, several imputation techniques will be considered based on the variables observed in the subject. In addition, the results obtained with and without the imputations will be compared to explore the effect of the missing values on the estimators. A sensitivity analysis will be performed if a high number of values for key variables are missing.

For the statistical analysis, generalized linear regression models will be used for repeated measurements (with identity link function and normal distribution for the continuous responses and Log link function with negative binomial distribution for count responses). This will take into account the correlation structure within each subject and the time-intervention interactions. The existence of random slopes and intercepts will be explored. All the models will be compared with Akaike models and the model hypotheses will be verified. All analyses will be performed with STATA 14.

ELIGIBILITY:
Inclusion Criteria:

* Belong to the group of neonates treated in neonatal intensive care units during the dates on which the sample will be taken.
* Clinical evaluation by the neonatologist indicating the infant's possible participation in the study.
* The neonate is between the gestational age of 28 and 37 weeks.

Exclusion Criteria:

* Mother is not able to give consent due to mental incapacity.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2017-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The Bayley-III Cognitive Scale | six month
  The Bayley III scales of infant development in English, based on which a metric scale will be used with a mean of 100 and a standard deviation of 15, and a range from 40-160, for the following subscales
The Bayley-III Motor Scale | six months
  The Bayley III scales of infant development in English, based on which a metric scale will be used with a mean of 100 and a standard deviation of 15, and a range from 40-160, for the following subscales
The Bayley-III Language Scale | six months
  The Bayley III scales of infant development in English, based on which a metric scale will be used with a mean of 100 and a standard deviation of 15, and a range from 40-160, for the following subscales
The Bayley-III Social-Emotional Scale | six months
  Composite score equivalents available in order to total the score of each subscale.
The Bayley-III Adaptive Behavior Scale | six months
  The scores of all the skill areas are combined to create the infant's global measurement scale for the subscale corresponding to Adaptive development.

SECONDARY OUTCOMES:
Heart rate | Everyday during all the follow-up period in neonatal intensive care unit (an average of 1 month). Also, it will be measured while neonate is receiving the intervention
Weight | Everyday during all the follow-up period in neonatal intensive care unit (an average of 1 month).
Blood pressure | Everyday during all the follow-up period in neonatal intensive care unit (an average of 1 month).. Also, it will be measured while neonate is receiving the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Manuela Beltran, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Diggle P, Heagerty P, Liang KY, Zeger S. Analysis of Longitudinal Data. Second edition. Oxford, UK: Oxford University Press, 2013.
- [Result] Loewy J. NICU music therapy: song of kin as critical lullaby in research and practice. Ann N Y Acad Sci. 2015 Mar;1337:178-85. doi: 10.1111/nyas.12648. PMID 25773633
- [Result] Standley JM, Cassidy J, Grant R, Cevasco A, Szuch C, Nguyen J, Walworth D, Procelli D, Jarred J, Adams K. The effect of music reinforcement for non-nutritive sucking on nipple feeding of premature infants. Pediatr Nurs. 2010 May-Jun;36(3):138-45. PMID 20687305
- [Result] Standley J. Music therapy research in the NICU: an updated meta-analysis. Neonatal Netw. 2012 Sep-Oct;31(5):311-6. doi: 10.1891/0730-0832.31.5.311. PMID 22908052
- [Result] Whitelaw A. Core Concepts: Intraventricular Hemorrhage NeoReviews 12 (2): e94-e10, 2011
- [Result] Auto FM, Amancio OM, Lanza FC. The effect of music on weight gain of preterm infants older than 32 weeks: a randomized clinical trial. Revista Paulista de Pediatria 33(4): e293-e299, 2015.
- [Result] Amini E, Rafiei P, Zarei K, Gohari M, Hamidi M. Effect of lullaby and classical music on physiologic stability of hospitalized preterm infants: a randomized trial. J Neonatal Perinatal Med. 2013 Jan 1;6(4):295-301. doi: 10.3233/NPM-1371313. PMID 24441085
- [Result] Lai HL, Chen CJ, Peng TC, Chang FM, Hsieh ML, Huang HY, Chang SC. Randomized controlled trial of music during kangaroo care on maternal state anxiety and preterm infants' responses. Int J Nurs Stud. 2006 Feb;43(2):139-46. doi: 10.1016/j.ijnurstu.2005.04.008. Epub 2005 Jul 5. PMID 15996669
- [Result] Macpherson H. Pragmatic clinical trials. Complement Ther Med. 2004 Jun-Sep;12(2-3):136-40. doi: 10.1016/j.ctim.2004.07.043. PMID 15561524
- [Result] Patsopoulos NA. A pragmatic view on pragmatic trials. Dialogues Clin Neurosci. 2011;13(2):217-24. doi: 10.31887/DCNS.2011.13.2/npatsopoulos. PMID 21842619